CLINICAL TRIAL: NCT06795646
Title: Clinical Classification and Prediction System of MAFLD Based on Liver Biopsy
Brief Title: Clinical Classification of MAFLD Based Liver Biopsy
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Fudan University (Other); Tianjin Second People's Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); The Affiliated Hospital of Hangzhou Normal University (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hong You, Vice-President, Beijing Friendship Hospital
Other Study IDs: 2023ZD0508702; 2023ZD0508702 (Other Grant/Funding Number: Noncommunicable Chronic Diseases-National Science and Technology Major Project)
Record Dates: First submitted 2025-01-20; First posted 2025-01-28 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Metabolic Dysfunction Associated Steatotic Liver Disease; Metabolic Dysfunction-associated Steatohepatitis (MASH)
Keywords: MAFLD; MASLD; liver-biopsy; classification; prediction model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — serum, PBMC, plasma, urine, feces, liver-biopsy tissues
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MAFLD diagnosed by liver-biopsy: retrospective and prospective cohort about MAFLD diagnosed by liver-biopsy

SUMMARY:
Metabolic dysfunction-associated Fatty Liver Disease (MAFLD), also known as Non-Alcoholic Fatty Liver Disease (NAFLD), is the most common chronic progressive liver disease in China. It is closely related to the high incidence of cardiovascular-renal-metabolic syndrome and both liver and non-liver malignancies, posing a serious threat to public health. However, the diagnostic criteria for MAFLD are not unified globally, and the classification and staging still rely on liver biopsy for pathological assessment. The characteristics, mechanisms, and predictive indicators of liver and extrahepatic disease outcomes in MAFLD patients are not yet clear.

The severe form of MAFLD, metabolic dysfunction-associated steatohepatitis (MASH), has been a hot and challenging area of research for non-invasive tests (NITs). However, serum markers, imaging examinations, and novel markers under development cannot replace liver biopsy for the diagnosis of MASH. Clinically, the disease outcomes of MAFLD mainly depend on metabolic cardiovascular risk factors and fibrosis staging. Both liver biopsy and NIT-diagnosed advanced fibrosis and cirrhosis can predict liver-related events and all-cause mortality risks in MAFLD patients. Artificial intelligence and machine learning methods can improve the consistency of pathologists in diagnosing MASH and fibrosis. The Agile score, which combines gender, T2DM status, AST/ALT ratio, platelet count, and liver stiffness measurement (LSM), can improve the diagnostic efficacy of advanced fibrosis and cirrhosis in MAFLD patients and the efficiency of predicting liver-related events. However, the predictive effect of fibrosis staging and its changes on liver cancer needs to be improved. There is a lack of high-quality research on early warning indicators for the incidence of CVD, chronic kidney disease, and non-liver malignancies in MAFLD patients. It is necessary to explore the role of conventional indicators such as low-density lipoprotein cholesterol, lipoprotein(a), uric acid, and high-sensitivity C-reactive protein, as well as multi-omics parameters, in the classification, staging, and risk prediction of MAFLD.

MAFLD is an increasingly serious public health issue associated with a higher risk of liver-related events, cardiovascular-renal-metabolic syndrome, and malignancies. The prevalence of MAFLD in China is high, but the rate of standardized management is low. Even patients with the same classification and staging often have different clinical characteristics and outcomes. There is currently a lack of a clinical classification and early warning system for MAFLD that combines metabolic cardiovascular risk factors and NITs for different outcome risks.

DETAILED DESCRIPTION:
1. Recruitment and Data Collection:

   On the basis of an existing cohort of 1,500 liver biopsy cases, recruit an additional 500 cases from a national multicenter liver biopsy follow-up cohort (totaling 2,000 cases). Collect demographic, anthropometric, laboratory, imaging, and liver biopsy results for these patients.

   Concurrently, biological samples, including blood, urine, feces, and liver biopsy tissues, will be collected. Utilize these samples to perform quantitative metabolite information based on database matching. Employ techniques such as genomics, epigenomics, proteomics, metabolomics, immunomics, and microbiome metagenomics to screen for differential biomarkers across different subgroups.

   Combine these findings with clinical and imaging parameters of MAFLD patients to analyze and explore key parameters and molecules at different stages and outcomes of MAFLD disease progression.
2. Development and Validation of a Diagnostic and Prognostic System:

Based on key molecules identified through multi-omics, in conjunction with characteristic parameters from clinical and imaging data of MAFLD patients, use machine learning methods (such as random forests neural networks) combined with logistic regression to establish a novel non-invasive diagnostic and prognostic assessment system for adverse outcomes (cardiovascular events, non-liver malignancies, and liver-related events).

Validate this new assessment system to ensure its reliability and accuracy in predicting disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound confirmation of fatty liver and the presence of at least one of the following metabolic cardiovascular risk factors:

  1. BMI ≥ 24 kg/m² or waist circumference ≥ 90 cm (men) and 85 cm (women) or excessive body fat content and body fat percentage.
  2. Fasting blood glucose ≥ 6.1 mmol/L or 2-hour post-load blood glucose ≥ 7.8 mmol/L or HbA1c ≥ 5.7% or history of Type 2 Diabetes Mellitus (T2DM) or Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) ≥ 2.5.
  3. Fasting serum triglycerides ≥ 1.70 mmol/L or currently receiving lipid-lowering drug therapy.
  4. Serum high-density lipoprotein cholesterol (HDL-C) ≤ 1.0 mmol/L (men) and 1.3 mmol/L (women) or currently receiving lipid-lowering drug therapy.
  5. Blood pressure ≥ 130/85 mmHg or currently receiving antihypertensive drug therapy.
* histology of liver-biopsy

Exclusion Criteria:

* Excessive Alcohol Consumption: Individuals who consume alcohol equivalent to ≥30 grams of ethanol per day for males, or ≥20 grams of ethanol per day for females, or those with missing alcohol consumption information.
* Viral Hepatitis Markers: Individuals who are positive for hepatitis B surface antigen (HBsAg), positive for hepatitis C virus (HCV) antibodies, or have missing information regarding these markers.
* History of Serious Medical Conditions: Individuals with a history of malignant tumors, cardiovascular diseases, chronic kidney disease, decompensated liver cirrhosis (manifested by ascites, gastrointestinal bleeding, hepatic encephalopathy, hepatorenal syndrome, etc.), or those who have undergone liver transplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MAFLD patients diagnosis by liver biopsy
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-02-08 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
composite endpoint | 1-20 years
  Number of participants with the composite endpoint, including
  A. Liver-Related Events:
  Cirrhosis Liver decompensation Hepatocellular carcinoma Liver transplantation
  B. Metabolic Diseases:
  Type 2 Diabetes Mellitus (T2DM) Hypertension Dyslipidemia Gout
  C. Cardiovascular Diseases (CVD):
  Coronary heart disease Stroke Heart failure Atrial fibrillation
  D. Non-Liver Malignancies:
  Colorectal adenoma/adenocarcinoma Gastric cancer Esophageal cancer Pancreatic cancer Gallbladder cancer Lung cancer Prostate cancer Hematological malignancies E. Chronic Kidney Disease
  F. Mortality:
  Liver disease-related deaths Cardiovascular disease-related deaths Other causes of death

SECONDARY OUTCOMES:
Liver-Related Events | 1-20 years
  Number of participants with liver-related events, including Cirrhosis, Liver decompensation, Hepatocellular carcinoma, Liver transplantation
Metabolic Diseases | 1-20 years
  Number of participants with metabolic disease, including Type 2 Diabetes Mellitus (T2DM), Hypertension, Dyslipidemia, Gout
Cardiovascular Diseases (CVD) | 1-20 years
  Number of participants with CVD, including Coronary heart disease, Stroke, Heart failure, Atrial fibrillation
Non-Liver Tumors | 1-20 years
  Number of participants with non-liver tumors, including colorectal adenoma/adenocarcinoma, gastric cancer, esophageal cancer, pancreatic cancer, gallbladder cancer, lung cancer, prostate cancer, hematological malignancies and so on
Chronic Kidney Disease | 1-20 years
  Number of participants with chronic kidney disease
Mortality | 1-20 years
  Number of participants including liver disease-related deaths, cardiovascular disease-related deaths, and Other causes of death

OTHER OUTCOMES:
biomarker by proteomics | baseline
  the clinical classification of MASLD by proteomics
biomarker by metabolomics | baseline
  the clinical classification of MASLD by metabolomics
biomarker by Immunomics | baseline
  the clinical classification of MASLD by immunomics
biomarker by Microbial Metagenomics | baseline
  the clinical classification of MASLD by microbial metagenomics

CONTACTS AND LOCATIONS:
Overall Officials: Hong You, PhD. / M.D., Principal Investigator — Beijing Friendship Hospital
Locations (6):
- China (6):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Xicheng
  - Hangzhou Normal University Affiliated Hospital, Hangzhou, Xicheng
  - Zhongshan Hospital, Fudan University, Shanghai, Xicheng
  - Shanghai Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Tianjin Second People's Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Patient Demographics, Anthropometrics, Serological, and Imaging Data, and Liver Biopsy Scores
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the project finished
Access Criteria: ask the principle investigator